CLINICAL TRIAL: NCT03725384
Title: Daily vs. Every Other Day Oral Iron Supplementation in Patients With Absolute Iron Deficiency Anemia (DEODO): a Multi-centered, Pilot Randomized Controlled Trial
Brief Title: Daily vs. Every Other Day Oral Iron Supplementation in Patients With Absolute Iron Deficiency Anemia
Acronym: DEODO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO ID 1534
Record Dates: First submitted 2018-10-23; First posted 2018-10-31 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-05

CONDITIONS: Anemia; Iron Deficiency Anemia
Keywords: Anemia; Iron deficiency; hemoglobin; oral iron; Ferrous sulfate
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferrous sulfate; Tablets; Iron; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous Sulfate and Vitamin C every other day (Experimental): Ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every other day for 12 weeks
  Interventions: Drug: Ferrous Sulfate 300Mg Tablet; Drug: Vitamin C 500Mg tablet
- Ferrous Sulfate and Vitamin C daily (Active Comparator): Ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every day for 12 weeks
  Interventions: Drug: Ferrous Sulfate 300Mg Tablet; Drug: Vitamin C 500Mg tablet

INTERVENTIONS:
Drug: Ferrous Sulfate 300Mg Tablet — oral dose of Ferrous Sulfate (300 mg) every day versus every other day along with vitamin C
  Other Names: Iron; Oral iron
Drug: Vitamin C 500Mg tablet — Vitamin C 500 Mg tablet every day versus every other day along with ferrous sulfate
  Other Names: Ascorbic acid

SUMMARY:
Iron deficiency anemia is a global health problem and the most common cause of anemia worldwide. Patients with iron deficiency (ID) and IDA can present with a multitude of symptoms including fatigue, restless legs syndrome and pica.Oral iron supplementation is associated with increasing hemoglobin in multiple studies in women, pregnant women and elderly patients.However, the optimal dose and frequency of oral iron supplementation for treatment remains unclear. The current proposed study attempts to address this gap in the literature.

DETAILED DESCRIPTION:
This is a pilot, pragmatic, non-inferiority, open label randomized controlled trial (RCT) in outpatients with iron deficiency anemia to evaluate the effectiveness of oral ferrous sulfate 300mg (60mg elemental iron) once daily versus every other day to improve hemoglobin at 12 weeks post-initiation. The rationale for this study includes: (1) IDA is a common and prevalent condition with potential adverse consequences if left untreated; (2) optimizing effectiveness of oral iron supplementation while minimizing side effects will improve treatment for patients.

Because IDA is a global health problem, common in clinical practice and treatable, this study will have a significant practical impact on how clinicians treat outpatients with iron deficiency anemia and how patients tolerate therapy.

For the patient, the expected benefit from taking part in this study is the potential to improve and treat iron deficiency anemia. These potential changes may lead to improved symptoms associated with iron deficiency anemia, such as cognitive and physical functioning, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years;
* Outpatients with iron deficiency anemia defined as Hb less than 120 g/L in women or 130g/L in men; AND ferritin less than 30 mcg/L

Exclusion Criteria:

* • Pregnancy

  * Currently breastfeeding
  * Known history of inflammatory bowel disease
  * Known history of celiac disease
  * Known history of thalassemia or thalassemia trait
  * Known inherited bleeding disorder
  * Known intolerance or lack of response to oral ferrous gluconate, sulfate or fumarate in the last 12 weeks
  * Multivitamin and mineral supplements (35 mg or more of elemental iron per day) in the 2 weeks prior to randomization
  * Allergy to oral iron
  * Allergy to any of the following medicinal and non-medicinal ingredients in ferrous sulfate: ferrous sulphate, calcium citrate, crospovidone, FD&C Red #40-Aluminum lake, FD&C Yellow #6-Aluminum Lake, magnesium stearate, microcrystalline cellulose, polyethylene glycol, polyvinyl alcohol, purified water, talc titanium dioxide
  * Allergy to any of the following medicinal and non-medicinal ingredients in vitamin C: Ascorbic acid, Colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, microcrystalline cellulose and stearic acid
  * Intravenous iron therapy in the past 12 weeks
  * On anticoagulant therapy (e.g. warfarin, apixaban, dabigatran, edoxaban, rivaroxaban) initiated in the past 6 months
  * Surgery planned in upcoming 12 weeks
  * Chemotherapy planned in upcoming 12 weeks
  * Blood donation planned in upcoming 12 weeks
  * Previously enrolled in the study
  * Creatinine clearance less than 30 mL/min
  * Hemoglobin less than 80 g/L with active bleeding (defined as WHO grade 2 bleeding or higher in the past week)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Yulia Lin, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Kron A, Del Giudice ME, Sholzberg M, Callum J, Cserti-Gazdewich C, Swarup V, Huang M, Distefano L, Anani W, Skeate R, Armali C, Lin Y. Daily versus every other day oral iron supplementation in patients with iron deficiency anemia (DEODO): study protocol for a phase 3 multicentered, pragmatic, open-label, pilot randomized controlled trial. Pilot Feasibility Stud. 2022 May 4;8(1):98. doi: 10.1186/s40814-022-01042-y. PMID 35509085
- [Background] Lin Y, Del Giudice ME, Kron A, Meirovich H, Sholzberg M, Swarup V, Huang M, Distefano L, Anani WQ, Armali C, Bussel JB, Callum J. A pilot feasibility trial of daily versus every other day oral iron supplementation in patients with iron deficiency anaemia. Br J Haematol. 2023 Jun;201(5):1000-1004. doi: 10.1111/bjh.18792. Epub 2023 Mar 31. No abstract available. PMID 36999886
- See also: Final manuscript - letter to the editor — https://pubmed.ncbi.nlm.nih.gov/36999886/
- See also: Study protocol — https://pubmed.ncbi.nlm.nih.gov/35509085/

RESULTS

PARTICIPANT FLOW:
Groups:
- Iron Daily: Ferrous sulfate (iron) 300mg tablet and vitamin C 500mg tablet taken by mouth every day for 12 weeks
- Iron Every Other Day: Ferrous sulfate (iron) 300mg tablet and vitamin C 500mg tablet taken by mouth every other day for 12 weeks
Period: Overall Study
Arm/Group | Iron Daily | Iron Every Other Day
Started | 24 | 27
Completed | 21 | 25
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Iron Every Other Day: Ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every other day for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (18.1) | 44.4 (17.1) | 45.7 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 27 | 51
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (6.7) | 27.0 (7.0) | 26.5 (6.8)
Reason for iron deficient anemia (IDA) diagnosis [Count of Participants; unit: Participants]
  Menorrhagia | 11 | 17 | 28
  Blood donation | 6 | 3 | 9
  Gastrointestinal | 4 | 4 | 8
  Other | 3 | 3 | 6
History of bleeding in the past 2 months [Count of Participants; unit: Participants] | 16 | 23 | 39
Menstrual bleeding, pictorial blood assessment chart >/= 100 [Count of Participants; unit: Participants] | 7 | 16 | 23
History of rheumatological disorders [Count of Participants; unit: Participants] | 4 | 3 | 7
Medication history [Count of Participants; unit: Participants]
  Ranitidine | 0 | 1 | 1
  Proton pump inhibitor | 1 | 0 | 1
Oral iron use in the past year [Count of Participants; unit: Participants] | 13 | 13 | 26
IV iron use in the past year [Count of Participants; unit: Participants] | 1 | 5 | 6
Baseline haemoglobin [Mean (Standard Deviation); unit: g/L] | 110 (13) | 110 (10) | 110 (11)
Baseline haemoglobin <100 g/L [Count of Participants; unit: Participants] | 3 | 3 | 6
Baseline mean corpuscular volume (MCV) [Mean (Standard Deviation); unit: fL] | 80.0 (8.2) | 80.6 (8.0) | 80.3 (8.1)
Baseline reticulocyte count [Median (Inter-Quartile Range); unit: x10^9 cells/L] | 48 [39 to 54] | 47 [41 to 65] | 48 [41 to 62]
Baseline ferritin [Median (Inter-Quartile Range); unit: mu grams/L] | 9 [5 to 17] | 9 [4 to 11] | 9 [4 to 14]
Baseline serum iron [Median (Inter-Quartile Range); unit: mu mol/L] | 8 [5 to 11] | 5 [4 to 9] | 7 [5 to 11]
Baseline C reactive protein [Median (Inter-Quartile Range); unit: mg/L] | 0.9 [0.6 to 2.0] | 1.0 [0.7 to 3.3] | 0.9 [0.6 to 3.0]
Baseline C reactive protein >/=5 mg/L [Count of Participants; unit: Participants] | 1 | 4 | 5
Baseline creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.83 [0.78 to 0.90] | 0.70 [0.64 to 0.89] | 0.78 [0.67 to 0.89]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrolling Patients in the Trial
Description: Enrollment in the trial will be defined as documentation of informed consent for patients approached. The primary outcome of this study is the feasibility of enrolling 52 participants in the trial over a 2-year period. Eligibility based on lab criteria was determined after consent.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Total Number Screened for Eligbility: Total number of participants screened for eligibility to be included in the study
Arm/Group | Total Number Screened for Eligbility
Number analyzed (Participants) | 216
participants | 85

2. Secondary Outcome: Proportion of Eligible Participants Consenting
Description: Proportion of eligible patients after initial inclusion/exclusion screening that consent to participating in the study. Eligibility based on lab criteria was determined after consent.
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Groups:
- Total Number Screened for Eligibility: Total number of patients who were screened for eligibility to be included in the trial
Arm/Group | Total Number Screened for Eligibility
Number analyzed (Participants) | 216
Proportion of participants | 0.39

3. Secondary Outcome: Proportion of Patients Receiving the Allocated Treatment
Description: Proportion of patients who signed informed consent and received the allocated treatment they were randomly assigned to.
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Groups:
- Total Number Allocated to Daily Iron: Total number of patients who were allocated to receive ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every day for 12 weeks
- Total Number Allocated to Iron Every Other Day: Total number of patients allocated to receive ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every other day for 12 weeks
- Total Number of Patients Allocated to Study Arms: Total number of patients that were allocated to one of the study arms
Arm/Group | Total Number Allocated to Daily Iron | Total Number Allocated to Iron Every Other Day | Total Number of Patients Allocated to Study Arms
Number analyzed (Participants) | 24 | 27 | 51
Proportion of participants | 0.96 | 1 | 0.98

4. Secondary Outcome: Proportion of Patients Completing Laboratory Tests
Description: Proportion of treated patients who completed both 4 week and 12 week laboratory tests
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Groups:
- Total Number Participants Receiving Daily Iron: Total number of participants who received daily iron during the study.
- Total Number Participants Receiving Iron Every Other Day: Total number of participants who received oral iron every other day during the study.
- Total Number Treated: Total number of patients who received either daily or every other day oral iron during the study.
Arm/Group | Total Number Participants Receiving Daily Iron | Total Number Participants Receiving Iron Every Other Day | Total Number Treated
Number analyzed (Participants) | 23 | 27 | 50
Proportion of participants | 0.91 | 0.81 | 0.86

5. Secondary Outcome: Proportion of Treated Patients Completing Side Effect Questionnaire at Week 4, 8 and 12
Description: Proportion of treated patients completing 4 week, 8 week and 12 week side effect questionnaire
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Groups:
- Iron Daily: Ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every day for 12 weeks
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 23 | 27
Proportion of participants | 0.91 | 0.85

6. Secondary Outcome: Proportion of Patients Completing FACIT-fatigue Scale
Description: Proportion of patients who received treatment and completed 4 week, 8 week and 12 week FACIT-fatigue scale
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 23 | 27
Proportion of participants | 0.91 | 0.89

7. Secondary Outcome: Adherence to Treatment
Description: Adherence was measured by the proportion of treated patients who took at least 90% of their prescribed doses
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 23 | 27
Proportion of participants | 0.78 | 0.82

8. Secondary Outcome: Proportion of Treated Patients Requiring a Step Down in Therapy
Description: Proportion of treated patients requiring a step down in therapy by Week 4 and Week 12 (same proportions at both time points).
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 24 | 27
Proportion of participants | 0.13 | 0

9. Secondary Outcome: Hemoglobin Increment
Description: Hemoglobin increment at 4 and 12 weeks is defined as the 4 or 12 week hemoglobin value minus the baseline hemoglobin value
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Iron Daily: Participants receiving oral iron on a daily basis
- Iron Every Other Day: Participants receiving oral iron every other day.
- Total: Includes participants in the daily iron group and every other day iron group.
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
g/L
  Hemoglobin at baseline | 110 (13) | 110 (10) | 110 (11)
  Hemoglobin at 4 weeks | 122 (7) | 119 (10) | 121 (9)
  Hemoglobin at 12 weeks | 131 (9) | 126 (8) | 129 (9)

10. Secondary Outcome: Proportion With Complete Hemoglobin Response
Description: Proportion with complete hemoglobin response defined as hemoglobin greater than or equal to 120 g/L in women; and 130 g/L in men at 4 weeks and 12 weeks
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Arm/Group | Ferrous Sulfate and Vitamin C Every Other Day | Ferrous Sulfate and Vitamin C Daily
Number analyzed (Participants) | 27 | 24
Proportion of participants | 0.59 | 0.75

11. Secondary Outcome: Reticulocyte Count
Description: Change in reticulocyte count at 4 and 12 weeks defined as the 4 or 12 week reticulocyte count minus the baseline reticulocyte count
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: x10^9 cells/ L
Groups:
- Iron Daily: Participants receiving oral iron daily.
- Total: Includes participants in the iron daily group and the iron every other day group.
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
x10^9 cells/ L
  Baseline reticulocyte count | 48 [39 to 54] | 47 [41 to 65] | 48 [41 to 62]
  Week 4 reticulocyte count | 61 [45 to 71] | 65 [48 to 79] | 64 [47 to 78]
  Week 12 reticulocyte count | 47 [39 to 56] | 52 [42 to 62] | 47 [41 to 61]

12. Secondary Outcome: Change in Ferritin at 12 Weeks
Description: Change in ferritin at 12 weeks, defined as the value at 12 weeks minus the baseline value.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
mcg/L
  Baseline ferritin | 9 [5 to 17] | 9 [4 to 11] | 9 [4 to 14]
  Week 12 ferritin | 30 [23 to 39] | 23 [20 to 34] | 27 [20 to 36]

13. Secondary Outcome: Change in Serum Iron at 12 Weeks
Description: Change in serum iron at 12 weeks defined as the value at 12 weeks minus the baseline value
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: micro mol/L
Groups:
- Total: Includes participants in iron daily group and iron every other day group.
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
micro mol/L
  Baseline serum iron | 8 [5 to 11] | 5 [4 to 9] | 7 [5 to 11]
  Week 12 serum iron | 17 [16 to 25] | 12 [9 to 16] | 16 [11 to 19]

14. Secondary Outcome: Change in TSAT at 12 Weeks
Description: Change in transferrin saturation (TSAT) at 12 weeks defined as the value at 12 weeks minus the baseline value. Interquartile range represents Q1 (25th percentile) to Q3 (75th percentile)
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
percentile
  Baseline TSAT | 11 [6 to 17] | 7 [6 to 10] | 9 [4 to 14]
  Week 12 TSAT | 26 [21 to 42] | 18 [14 to 27] | 23 [16 to 31]

15. Secondary Outcome: FACIT-fatigue Score at 4, 8 and 12 Weeks
Description: Quality of life (FACIT-fatigue scale) at 4, 8 and 12 weeks. Functional Assessment of Chronic Illness Therapy (FACIT) - fatigue scale.
  On this scale, lower scores indicate better symptoms and higher scores represent worse symptoms. The FACIT-fatigue scale has a range from 0 to 52.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Total/All Participants: Overall FACIT-Fatigue Scale at weeks 4, 8, and 12.
Arm/Group | Iron Daily | Iron Every Other Day | Total/All Participants
Number analyzed (Participants) | 24 | 27 | 51
score on a scale
  Week 4 FACIT-fatigue score | 23.9 (9.8) | 26.3 (9.7) | 25.2 (9.7)
  Week 8 FACIT-fatigue score | 21.5 (8.5) | 24.9 (11.4) | 23.4 (10.2)
  Week 12 FACIT-fatigue score | 20.1 (8.5) | 21.9 (9.9) | 21.0 (9.3)

16. Secondary Outcome: Proportion of Patients With Side Effects at 4, 8 and 12 Weeks
Description: Proportion of patients with side effects at 4, 8 and 12 weeks, as determined by the oral iron side effect questionnaire
Time Frame: 12 weeks
Measure: Number; unit: Proportion of participants
Groups:
- Total/All Participants: Overall proportion of patients with adverse effects.
Arm/Group | Iron Daily | Iron Every Other Day | Total/All Participants
Number analyzed (Participants) | 24 | 27 | 51
Proportion of participants
  Week 4 | 0.38 | 0.56 | 0.47
  Week 8 | 0.33 | 0.48 | 0.41
  Week 12 | 0.33 | 0.44 | 0.39

17. Secondary Outcome: Proportion of Patients Who Stopped Oral Iron Due to Side Effects
Description: Number of patients who discontinued oral iron therapy due to side effects by week 12.
Time Frame: 12 weeks
Measure: Number; unit: Proportion of participants
Arm/Group | Iron Daily | Iron Every Other Day | Total
Number analyzed (Participants) | 24 | 27 | 51
Proportion of participants | 0 | 0 | 0

18. Secondary Outcome: Number of Patients in Need of Escalation Therapy
Description: Need for escalation in therapy (increase in oral iron regimen from every other day to daily, need for intravenous iron, need for transfusion, visit to emergency department related to anemia) assessed at 12 weeks
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 24 | 27
Participants | 0 | 0

19. Secondary Outcome: Proportion of Patients With a Drop in Hemoglobin at Weeks 4 and 12
Description: Proportion of patients with a drop in hemoglobin of 10 g/L or more at weeks 4 and 12
Time Frame: 2 years
Measure: Number; unit: Proportion of participants
Groups:
- Iron Every Other Day: Ferrous sulfate 300mg tablet and vitamin C 500mg tablet taken by mouth every other day for 12 weeks
  Ferrous Sulfate 300Mg Tablet: oral dose of Ferrous Sulfate (300 mg) every day versus every other day along with vitamin C
  Vitamin C 500Mg tablet: Vitamin C 500 Mg tablet every day versus every other day along with ferrous sulfate
Arm/Group | Iron Daily | Iron Every Other Day
Number analyzed (Participants) | 24 | 27
Proportion of participants | 0 | 0

20. Secondary Outcome: Types of Adverse Effects at 4 Weeks
Description: Proportion of patients with each type of adverse event at week 4.
Time Frame: 4 Weeks
Measure: Number; unit: Proportion of participants
Groups:
- Total/All Participants: Overall proportion of patients with the adverse effect.
Arm/Group | Iron Daily | Iron Every Other Day | Total/All Participants
Number analyzed (Participants) | 24 | 27 | 51
Proportion of participants
  Constipation | 0.25 | 0.22 | 0.24
  Nausea | 0.17 | 0.26 | 0.22
  Headache | 0.17 | 0.26 | 0.22
  Breathlessness | 0.17 | 0.26 | 0.22
  Heartburn | 0.08 | 0.30 | 0.20
  Abdominal pain | 0.08 | 0.19 | 0.14
  Diarrhea | 0.08 | 0.19 | 0.14
  Vomiting | 0.04 | 0.11 | 0.08
  Other | 0.21 | 0.22 | 0.22

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at weeks 4, 8, and 12.
Description: Adverse events were documented at each follow-up according to the Common Terminology Criteria for Adverse Events (Version 5.0). A modified adverse effects of oral iron questionnaire was used.
Arm/Group | Ferrous Sulfate and Vitamin C Every Other Day | Ferrous Sulfate and Vitamin C Daily | Total/All Participants
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/51
Other Adverse Events (participants affected / at risk) | 15/27 | 9/24 | 24/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferrous Sulfate and Vitamin C Every Other Day (N=27) | Ferrous Sulfate and Vitamin C Daily (N=24) | Total/All Participants (N=51)
Constipation (Gastrointestinal disorders) | 6 | 6 | 12 — Adverse effect reported at week 4 using adverse effect questionnaire.
Nausea (Gastrointestinal disorders) | 7 | 4 | 11 — Adverse effect reported at week 4 using questionnaire
Headache (Nervous system disorders) | 7 | 4 | 11 — Adverse effect reported at Week 4 using questionnaire
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 11 — Adverse effect reported at week 4 using questionnaire
Heartburn (Gastrointestinal disorders) | 8 | 2 | 10 — Adverse effect reported at week 4 using questionnaire
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 7 — Adverse effect reported at week 4 using questionnaire
Diarrhea (Gastrointestinal disorders) | 5 | 2 | 7 — Adverse effect reported at week 4 using questionnaire
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 — Adverse effect reported at week 4 using questionnaire

LIMITATIONS AND CAVEATS:
The exclusion of previously intolerant oral iron patients may bias the study group. Slight imbalances in IDA cause between daily and EOD groups may favour hemoglobin improvement in the daily group. Lack of blinding could impact patient reporting on FACIT-fatigue or adverse effects. Using oral vitamin C may now be unnecessary; recent study shows no added benefit when it is taken with oral iron. The timing of the iron indices (serum iron, transferrin saturation) was not recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT03725384/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT03725384/ICF_001.pdf